CLINICAL TRIAL: NCT01697709
Title: Quetiapine Pharmacotherapy for Cannabis Dependence
Acronym: QUEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John Mariani MD, research psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6623; 1R01DA031826 (NIH)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Cannabis Dependence
Keywords: cannabis; marijuana; pharmacotherapy
MeSH Terms: conditions — Marijuana Abuse | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo medication
  Interventions: Drug: Placebo
- quetiapine (Experimental): Quetiapine treatment
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Quetiapine pharmacotherapy for cannabis dependence
  Other Names: Seroquel
  Arms: quetiapine
Drug: Placebo — placebo capsules
  Other Names: Matched Placebo
  Arms: Placebo

SUMMARY:
Despite a benign public perception, marijuana use disorders represent a significant public health problem. The development of safe and effective pharmacotherapies for marijuana dependence is an important unmet public health need. Quetiapine, an effective atypical antipsychotic that acts by blocking serotonin type 2A, dopamine type 2, histamine type 1, and adrenergic receptors, is a promising treatment for substance use disorders. In animal models, quetiapine blocks the enhancement of reward by cocaine, which is likely due to its actions on both dopamine and non-dopamine neurotransmission. Clinical studies of quetiapine have shown benefit for the treatment of alcohol and cocaine use disorders.

Conceptually, the clinically prominent effects of quetiapine, namely sedation, anxiolysis, mood stabilization and appetite stimulation, are a good match for the symptoms of marijuana withdrawal. Most importantly, an open-label dose-finding study of quetiapine for the treatment of marijuana dependence conducted by our research group determined that quetiapine was well-tolerated and associated with reductions in marijuana use indicating that it is a promising agent deserving of further study in marijuana-dependent outpatients.

The proposed research project is a randomized double-blind placebo-controlled clinical trial to evaluate the efficacy of quetiapine for the treatment of marijuana dependence over a 12-week period. All participants will receive Medical Management, a medication adherence focused psychosocial intervention that facilitates compliance with study medication and other study procedures, promotes abstinence from marijuana and other substances, and encourages mutual-support group attendance. All participants will receive voucher incentives for compliance with study visit attendance, returning study medication bottles, and completing other study procedures, with the objective of achieving a highly compliant sample. The goal of this phase II clinical trial is to build on our promising open-label pilot study results and examine the efficacy of quetiapine on participants' marijuana consumption under placebo-controlled double-blind conditions using an abstinence-initiation model, where participants will be using marijuana regularly at study entry, reduce their use, and then achieve abstinence. The specific aims of the projects are to determine whether quetiapine is superior to placebo in 1) reducing marijuana use and 2) achieving abstinence.

DETAILED DESCRIPTION:
In a 12-week randomized double-blind placebo-controlled clinical trial, we will evaluate the efficacy of quetiapine for the treatment of marijuana dependence in 150 outpatients. Participants will be randomly assigned to treatment under double-blind conditions with either a fixed dosing schedule of quetiapine or placebo. All participants will receive Medical Management, a medication adherence focused psychosocial intervention that facilitates compliance with study medication and other study procedures, and promotes abstinence from marijuana and other substances. All participants will receive progressive voucher incentives for compliance with study visit attendance and completing other study procedures, with the objective of achieving a highly compliant sample.

The results of a dose-finding pilot study of quetiapine for the treatment of marijuana dependence (see Preliminary Studies) suggests that the ideal dosing for the proposed project is a single 300 mg dose every evening, achieved after a gradual three-week titration. Clinical experience with this medication for treatment of marijuana dependence indicates that a gradual upward titration of dose is advisable to maximize tolerability and that morning dosing was poorly tolerated. Quetiapine (immediate release formulation) will be administered in 25 and 100 mg capsules; placebo capsules will appear identical to the quetiapine capsules. Participants in both treatment arms will take the same number of pills on the same schedule. Study medication will be dispensed on a weekly basis starting with the baseline visit. Quetiapine will be titrated over a three-week period to the target dose of 300 mg or the maximum tolerated dose. The research psychiatrist will make dose reductions for tolerability if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV-TR criteria for current marijuana dependence
2. Reports using marijuana an average of 5 days per week over the past 28 days
3. Between the ages of 18 and 60
4. Able to provide informed consent and comply with study procedures
5. Seeking treatment for cannabis dependence

Exclusion Criteria:

1. Lifetime DSM-IV diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder.
2. Current DSM-IV criteria for any other psychiatric disorder that may, according to investigator's judgment, require either pharmacological or non-pharmacological intervention over the course of the study.
3. Patients prescribed psychotropic medications.
4. History of allergic reaction, intolerance, or hypersensitivity to Quetiapine.
5. Pregnancy, lactation, or failure to use adequate contraceptive methods in female patients who are currently engaging in sexual activity with men.
6. Unstable medical conditions, such as poorly controlled hypertension which might make participation hazardous.
7. Diabetes (whether controlled or not), meeting criteria for metabolic syndrome as defined by the NCEP (any 3 of the following: a. obesity [waist circumference > 40 inches], b. hyperglycemia [fasting glucose > 100 mg/dl or Rx], c. dyslipidemia [TG > 150 mg/dl or Rx], d. dyslipidemia [HDL cholesterol; 40 mg/dl (male), 50 mg/dl (female) or Rx], e. hypertension [130 mmHg systolic or > 85 mmHg diastolic or Rx]. Participants with a BMI > 35 will be excluded.
8. Current DSM-IV diagnosis of an alcohol or substance use disorder (abuse or dependence) other than marijuana or nicotine dependence.
9. Positive confirmed result on urine toxicology screen.
10. Are legally mandated to participate in a substance use disorder treatment program.
11. Increased risk for suicide.
12. QTc prolongation (screening electrocardiogram with Qtc > 450 msec for men, QTc > 470 msec for women) or history of QTc prolongation or using concomitant medications which prolong QTc interval.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Mariani, MD, Principal Investigator — Columbia University/NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study web site — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomized to one of the treatment arms at time of enrollment
Period: Overall Study
Arm/Group | Placebo | Quetiapine
Started | 64 | 66
Completed | 34 | 38
Not Completed | 30 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Quetiapine | Total
Number analyzed (Participants) | 64 | 66 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (8.7) | 32.7 (9.5) | 32.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 50 | 52 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 32
  Not Hispanic or Latino | 49 | 49 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 24 | 56
  White | 18 | 25 | 43
  More than one race | 3 | 8 | 11
  Unknown or Not Reported | 8 | 8 | 16
mood/anxiety disorder [Count of Participants; unit: Participants] | 14 | 14 | 28
Marijuana using days past 28 days [Mean (Standard Deviation); unit: days] | 26.8 (2.1) | 26.4 (2.5) | 26.6 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Marijuana Use, Daily Dollar Averaged Over 7 Days During Each of 12 Weeks of Study
Description: The median daily dollar value of marijuana used averaged over a one-week period for each of the 12 weeks as recorded by the Timeline Followback method
Time Frame: 12 weeks or length of participants involvement
Measure: Median (Inter-Quartile Range); unit: dollars
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 64 | 66
dollars
  week 1 | 14.00 [5.42 to 21.25] | 7.00 [3.18 to 12.86]
  week 2 | 10.00 [2.86 to 22.00] | 8.00 [3.02 to 12.70]
  week 3 | 7.14 [2.64 to 17.69] | 5.86 [3.29 to 11.61]
  week 4 | 6.43 [1.61 to 16.25] | 5.71 [2.57 to 12.00]
  week 5 | 6.43 [1.07 to 17.86] | 4.29 [1.43 to 9.29]
  week 6 | 5.71 [0.96 to 13.82] | 4.11 [1.32 to 9.79]
  week 7 | 3.70 [1.03 to 12.59] | 3.57 [1.43 to 7.52]
  week 8 | 2.86 [1.12 to 12.26] | 3.43 [1.18 to 6.00]
  week 9 | 6.43 [1.03 to 11.96] | 3.00 [1.43 to 7.00]
  week 10 | 5.35 [0.00 to 12.32] | 2.86 [0.29 to 5.14]
  week 11 | 3.21 [0.00 to 11.79] | 2.86 [0.00 to 5.14]
  week 12 | 1.00 [0.00 to 12.29] | 2.14 [0.00 to 5.25]

2. Primary Outcome: Number of Participants Stratified by Marijuana Abstinence Days Per Week
Description: The number of abstinent days per week over the 12 weeks of study as recorded by the Timeline Followback method. High Use group defined as 0-2 abstinent days per week, Medium Use Group as 3-5 abstinent days per week and Low Use Group as 6-7 abstinent days per week.
Time Frame: 12 weeks or length of participation
Population: participants were included in the weekly analysis who were still active in the trial at each given week.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 64 | 66
Participants
  Week 1: number analyzed (Participants) | 54 | 59
  Week 1: high use | 5 | 4
  Week 1: medium use | 9 | 9
  Week 1: low use | 40 | 46
  Week 2: number analyzed (Participants) | 49 | 55
  Week 2: high use | 8 | 4
  Week 2: medium use | 7 | 7
  Week 2: low use | 34 | 44
  Week 3: number analyzed (Participants) | 42 | 52
  Week 3: high use | 9 | 5
  Week 3: medium use | 5 | 14
  Week 3: low use | 28 | 33
  Week 4: number analyzed (Participants) | 40 | 49
  Week 4: high use | 8 | 8
  Week 4: medium use | 9 | 15
  Week 4: low use | 23 | 26
  Week 5: number analyzed (Participants) | 39 | 47
  Week 5: high use | 10 | 10
  Week 5: medium use | 7 | 16
  Week 5: low use | 22 | 21
  Week 6: number analyzed (Participants) | 39 | 46
  Week 6: high use | 13 | 10
  Week 6: medium use | 4 | 13
  Week 6: low use | 22 | 23
  Week 7: number analyzed (Participants) | 38 | 43
  Week 7: high use | 12 | 11
  Week 7: medium use | 9 | 15
  Week 7: low use | 17 | 17
  Week 8: number analyzed (Participants) | 38 | 43
  Week 8: high use | 12 | 10
  Week 8: medium use | 9 | 16
  Week 8: low use | 17 | 17
  Week 9: number analyzed (Participants) | 38 | 43
  Week 9: high use | 13 | 13
  Week 9: medium use | 7 | 15
  Week 9: low use | 18 | 15
  Week 10: number analyzed (Participants) | 36 | 41
  Week 10: high use | 14 | 13
  Week 10: medium use | 5 | 13
  Week 10: low use | 17 | 15
  Week 11: number analyzed (Participants) | 36 | 37
  Week 11: high use | 15 | 14
  Week 11: medium use | 5 | 12
  Week 11: low use | 16 | 11
  Week 12: number analyzed (Participants) | 34 | 37
  Week 12: high use | 17 | 15
  Week 12: medium use | 3 | 11
  Week 12: low use | 14 | 11

ADVERSE EVENTS:
Time Frame: over 12 weeks of study or length of participation
Arm/Group | Placebo | Quetiapine
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/66
Other Adverse Events (participants affected / at risk) | 34/64 | 46/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Quetiapine (N=66)
Hypertension (Cardiac disorders) | 24 (24) | 36 (36) — >130 or > 85
Hyperglycemia (General disorders) | 15 (15) | 18 (18) — >100 mg
Dyslipidemia (Endocrine disorders) | 11 (11) | 10 (10) — TG >150mg
drowsiness (General disorders) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/09/NCT01697709/Prot_000.pdf
  • Statistical Analysis Plan (2011-11-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT01697709/SAP_001.pdf